CLINICAL TRIAL: NCT02546843
Title: Deep Neuromuscular Blockade During Laparoscopic Surgery in Pediatric Patient and the Impact of the Depth of the Blockade on the Surgery Conditions, Perioperative Complications and Surgeon Satisfaction
Brief Title: Depth of Neuromuscular Blockade and the Perioperative Conditions in Laparoscopic Surgery in Pediatric Population
Acronym: PedLapBlock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Collaborators: KDCHOT FN Brno (Unknown)
Responsible Party: Principal Investigator, Petr Štourač, MD, MD,Ph.D, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KDAR FN Brno
Record Dates: First submitted 2015-09-05; First posted 2015-09-11 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Neuromuscular Blockade
Keywords: rocuronium; sugammadex; pediatric anesthesia; cisatracurium; surgical conditions
MeSH Terms: interventions — Rocuronium; cisatracurium; Neuromuscular Blockade

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): After anesthesia induction: intravenous cannulation, preoxygenation, sufentanil 0.2 μg/kg intravenously, propofol 2.0mg/kg the neuromuscular blockade will be induced with rocuronium 0.6 mg/kg (1 mg/kg only in a case of a rapid sequence induction).
  maintaining the depth of neuromuscular blockade - rocuronium: the appropriate depth of the block will be maintained with repeated boluses of rocuronium 0.3 mg/kg according to TOF 0, PTC 0-1.
  Specific Neuromuscular Blockade reversal will be performed with Sugammadex intravenously. The proper dosage of sugammadex will depend on the depth of the blockade:at TOF -1-2 (train-of-four) 2m g/kg, if TOF 0 and PTC(post-tetanic count) 0-1 4mg/kg of sugammadex will be administered
  Interventions: Drug: Rocuronium; Drug: Specific Neuromuscular Blockade reversal; Drug: maintaining the depth of neuromuscular blockade - rocuronium
- Group B (Active Comparator): After anesthesia induction: intravenous cannulation, preoxygenation, sufentanil 0.2 μg/kg intravenously, propofol 2.0mg/kg the neuromuscular blockade will be induced with cisatracurium 0.15mg/kg intravenously.
  Maintaining the depth of neuromuscular blockade - cisatracurium:the appropriate depth of the block will be maintained with repeated boluses of cisatracurium 0.03 mg/kg - according to TOF maintaining of muscular relaxation TOF 1.
  Nonspecific Neuromuscular Blockade reversal will be performed with neostigmine 0.03 mg/kg and atropine 0.02 mg/kg intravenously, the reversal will be applicated in case of TOF 1 or higher.
  Interventions: Drug: Cisatracurium; Drug: Nonspecific Neuromuscular Blockade reversal; Drug: maintaining the depth of neuromuscular blockade - cisatracurium

INTERVENTIONS:
Drug: Rocuronium — rocuronium 0.6 mg/kg intravenously (1 mg/kg only in a case of a rapid sequence induction)
  Other Names: Esmeron
  Arms: Group A
Drug: Cisatracurium — cisatracurium 0.15mg/kg intravenously
  Other Names: Nimbex
  Arms: Group B
Drug: Nonspecific Neuromuscular Blockade reversal — neostigmine 0.03 mg/kg and atropine 0.02 mg/kg intravenously
  Arms: Group B
Drug: Specific Neuromuscular Blockade reversal — Sugammadex intravenously aimed to reverse the neuromuscular blockade.According to neuromuscular blockade monitoring: at TOF - (train-of-four) 2m g/kg, if TOF 0 and PTC(post-tetanic count) 0-1 4mg/kg of sugammadex will be administered
  Arms: Group A
Drug: maintaining the depth of neuromuscular blockade - rocuronium — repeated boluses of rocuronium 0.3 mg/kg will be administered to maintain the muscular blockage - according to TOF 0, PTC 0-1
  Other Names: neuromuscular blockade
  Arms: Group A
Drug: maintaining the depth of neuromuscular blockade - cisatracurium — repeated boluses of cisatracurium 0.03 mg/kg will be administered to maintain the muscular blockage - according to TOFmaintaining of muscular relaxation TOF 1
  Other Names: neuromuscular blockade
  Arms: Group B

SUMMARY:
This randomized study prospectively evaluates our experience with administration of cisatracurium and rocuronium antagonized by sugammadex and evaluates the effects of various depths of neuromuscular blockage on providing optimal surgical conditions during laparoscopy with low-pressure capnoperitoneum.

DETAILED DESCRIPTION:
This randomized study prospectively evaluates our experience with administration of cisatracurium and rocuronium antagonized by sugammadex and evaluates the effects of various depths of neuromuscular blockage on providing optimal surgical conditions during laparoscopy with low-pressure capnoperitoneum.

After meeting inclusion criteria the patients will be randomized - - use of opaque envelopes, randomization into groups A and B in an operating theatre, study blinded for the patient (or his/her legal guardian) and surgeon.

Group A - muscle relaxation using rocuronium followed by sugammadex reversal (in a dose according to TOF - (train-of-four) 2-4mg/kg), depth of muscle relaxation TOF 0 PTC (post-tetanic count) 0-1 Group B - muscle relaxation using cisatracurium followed by decurarization (neostigmine 0.03 mg/kg and atropine 0.02 mg/kg)

Anesthesia management:

* intravenous cannulation, preoxygenation, sufentanil 0.2 μg/kg intravenously, propofol 2.0mg/kg and in Group A - rocuronium 0.6 mg/kg (1 mg/kg only in a case of a rapid sequence induction), in Group B - cisatracurium 0.15mg/kg
* orotracheal intubation, combined anesthesia using sevoflurane - MAC (minimal alveolar concentration) 1.0 with respect to the age of the patient
* ventilation: PCV (pressure-controlled ventilation ), PEEP (positive end-expiratory pressure) +5 cm H2O (aqua), normocapnia, FiO2 (fraction of inspired oxygen ) 1.0 until the intubation, afterwards 0.4 + AIR
* nasogastric tube placement

Management of neuromuscular blockade:

Group A - maintaining of deep muscular blockage - according to TOF 0, PTC 0-1, boluses of rocuronium 0.3 mg/kg are allowed Group B - maintaining of muscular relaxation TOF 1, boluses of cisatracurium 0.03 mg/kg are allowed Laparoscopy - capnoperitoneum pressure - 10 mmHg with a reduction to 8 mmHg if possible

During the surgery the surgical conditions will be scored by using Surgical scoring system: (1-2 surgeons involved):

1. Optimal conditions: there is a wide laparoscopic field, no movements or contractions
2. Good conditions: there is a wide laparoscopic field with singular movements or muscle contractions
3. Acceptable conditions: there is a wide laparoscopic field but muscle contractions and/or movements occur regularly. Additional neuromuscular blocking agent is required.
4. Poor conditions: the same as in grade 3 and in addition, there is a hazard of tissue damage.
5. Extremely poor conditions: the surgeon cannot work because of weak muscle relaxation, the patient is coughing. Additional neuromuscular blocking agent is essential.

Recovery from anesthesia:

* extubation - TOF 0.9 - using sugammadex in Group A (2-4 mg/kg according to the depth of muscle relaxation) or decurarization in Group B (atropine 0.02 mg/kg and neostigmine 0.03mg/kg)
* after standard 2-hour monitoring in the recovery room (heart rate, blood pressure, SpO2 (oxygen saturation by pulse oximetry), level of consciousness, PONV), patients will be observed in the intensive care unit for at least 24 hours Statistical analysis: (provided by IBA MUNI - Institute of biostatistic and analyses by Masaryk University Brno, Czech Republic)
* demographic parameters - age, gender, type and duration of surgery
* induction to general anesthesia - time until intubation (recognition of the capnogram curve)
* ventilation - changes in the inspiratory pressure during capnoperitoneum, increase of EtCO2 (end-tidal CO2)
* capnoperitoneal pressure
* surgical scoring system

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients aged 2 to 17 years (+ 364 days) eligible for laparoscopy (diagnostic laparoscopy, appendectomy, cholecystectomy, nephrectomy, splenectomy, tumor biopsy, varicocele correction, testicular retention)
* fasting of at least 6 hours
* ASA (American Society of Anesthesiology score) score 1 or 2
* signed informed consent of the legal guardian of the patient

Exclusion Criteria:

* disagreement of the patient or his/her legal guardian
* serious comorbidities - renal or hepatic disorders
* ASA score ≥ 3

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2015-12; Primary Completion 2018-09 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Surgical scoring system | intraoperatively
  During the surgery the blinded surgeon will grade surgical conditions due to surgical scoring system

SECONDARY OUTCOMES:
Number of adverse events | intraoperatively
  The adverse events will be monitored

CONTACTS AND LOCATIONS:
Overall Officials: Petr Štourač, MD, Ph.D, Study Chair — KDAR FN Brno
Locations (1):
- University Hospital Brno - FN Brno, Brno, Czech Republic, Czechia